CLINICAL TRIAL: NCT06585410
Title: A Phase 3 Randomized Study of Intralesional Cemiplimab Versus Primary Surgery in Participants With Early Stage Cutaneous Squamous Cell Carcinoma (CSCC)
Brief Title: Study of Intralesional Cemiplimab in Adult Patients With Early Stage Cutaneous Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-2251; 2024-511812-26-00 (Registry Identifier: EUCT Number)
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cutaneous Squamous Cell Carcinoma (CSCC)
Keywords: Dermato-Oncology; Cemiplimab; Early Stage; Skin Cancer; Non-Melanoma Skin Cancer; UV Skin Damage; Chronic Sun Exposure
MeSH Terms: conditions — Skin Neoplasms | interventions — cemiplimab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Investigational treatment
  Interventions: Drug: Cemiplimab
- Control Arm (Other): Standard of care treatment
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Drug: Cemiplimab — Administered per protocol
  Other Names: Libtayo
  Arms: Experimental Arm
Procedure: Standard of care — Primary surgery
  Arms: Control Arm

SUMMARY:
This study will test a study drug called cemiplimab to see if it can help treat early-stage cutaneous squamous cell carcinoma (CSCC), a type of skin cancer. Cemiplimab works by helping the immune system to kill cancer cells. It binds to a protein called programmed cell death-1 (PD-1) on the surface of certain immune cells.

The main purpose of this study is to compare how well cemiplimab works compared to surgery, when injected into the lesion.

The study is looking at:

* The side effects cemiplimab might cause
* How well cemiplimab works

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants who have a histologically confirmed invasive CSCC TL, as described in the protocol
2. Participants who have CSCC TL ≥1 cm and ≤2.0 cm (longest diameter) located in either the Head or Neck (HN), hand, or pre-tibial surface, as described in the protocol
3. Participants who are judged to be eligible for surgical resection of their CSCC TL and the method of planned surgical resection would be Micrographically oriented histographic surgery (Mohs) or other surgical method of Complete Margin Assessment (CMA). Participants for whom the planned surgery is surgical excision without margin control are not eligible
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1
5. Adequate hepatic, renal and bone marrow functions, as described in the protocol

Key Exclusion Criteria:

1. Participant in which the TL is a keratoacanthoma (KA), adenosquamous carcinoma, desmoplastic carcinoma, basal cell carcinoma, basosquamous.carcinoma, Bowen's disease, or CSCC in situ without an invasive component. (Note: For participants with invasive CSCC with a minor basaloid component, the patient may be eligible after discussion with the sponsor medical director.)
2. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for Immune-mediated Adverse Events (imAEs), as described in the protocol
3. History of non-infectious pneumonitis within the last 5 years
4. TL (lesion planned for intralesional therapy) or other non-target CSCC lesion in dry red lip (vermillion), oral cavity, or nasal mucosa

NOTE: Other protocol defined inclusion / exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2030-05-03 (Estimated); Study Completion 2030-05-03 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) as assessed by the investigator | Up to 1 year
EFS as assessed by the investigator | Up to 3 years

SECONDARY OUTCOMES:
Composite Complete Response (CCR) for Target Lesion (TL) | At week 13
  Experimental Arm
Non-Target Lesions (NTLs) in the Region of the Target Lesion (ROTL) | Baseline and at week 13
  Experimental Arm
Incidence of Treatment Emergent Adverse Events (TEAEs) | Up to 3 years
Severity of TEAEs | Up to 3 years
Size of surgical defect | At week 13
Size of biopsy defect | At week 13

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (48):
- United States (43):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Arkansas Research Trials, North Little Rock, Arkansas
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Stanford University, Redwood City, California
  - Peak Dermatology, Aesthetics and Wellness, Visalia, California
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Life Clinical Trials, Coral Springs, Florida
  - Dermatology Associates of the Palm Beaches, Delray Beach, Florida
  - University of South Florida, St. Petersburg, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Oak Dermatology, Naperville, Illinois
  - Dawes Fretzin Clinical Research - Shadeland Ave., Indianapolis, Indiana
  - Equity Medical, LLC, Bowling Green, Kentucky
  - US Dermatology Partners DBA DermAssociates, PC, Rockville, Maryland
  - Northeast Dermatology Associates, Beverly, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - MyMichigan Dermatologic Oncology, Midland, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Dermatology and Skin Cancer Center, Lee's Summit, Missouri
  - Washington University in St. Louis - Center for Dermatologic and Cosmetic Surgery, St Louis, Missouri
  - Las Vegas Dermatology, Las Vegas, Nevada
  - Metropolitan Dermatology, Clark, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Medical Center - Herbert Irving Center for Dermatology and Skin Cancer - Herbert Irving Pavilion, New York, New York
  - Rochester Dermatologic Surgery, P.C., Victor, New York
  - UNC Hospitals Dermatology and Skin Cancer Center at Southern Village, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Buckeye Dermatology - Springfield Office, Springfield, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Dermatology Health Specialists, Bend, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - The University of Texas at Austin Dell Medical School Ascension Medical Group, Austin, Texas
  - Reveal Research Institute, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Epiphany Dermatology, Lewisville, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - University of Utah Hospital, Salt Lake City, Utah
- Australia (5):
  - The Skin Hospital, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Dermatology Institute of Victoria (DIV), South Yarra, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has :
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * has the legal authority to share the data, and
  * has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: Clear — https://clear-clinicalstudy.com/en-us/